CLINICAL TRIAL: NCT04994327
Title: Bread Replacement - Facing the Challenge to Improve Its Quality for Better Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Paderborn University (Other); University of Leipzig (Other); Chalmers University of Technology (Other); Nofima (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 727565
Record Dates: First submitted 2021-07-07; First posted 2021-08-06 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Bread; Hyperglycemia; Glycemic Control; PreDiabetes
Keywords: beta-glucan; hyperglycemia; pre-diabetes
MeSH Terms: conditions — Hyperglycemia; Prediabetic State; Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: Multicenter
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-glucan bread (Experimental): Frozen bread is administered to the participants for home storage. Bread is thawed at home before consumption. Dosage: At least 3 slices of bread 6 days per week for 16 weeks
  Interventions: Other: Beta-glucan bread
- Control bread (Placebo Comparator): Frozen bread is administered to the participants for home storage. Bread is thawed at home before consumption. Dosage: At least 3 slices of bread 6 days per week for 16 weeks
  Interventions: Other: Beta-glucan bread

INTERVENTIONS:
Other: Beta-glucan bread — Frozen bread is administered to the participants for home storage. Bread is thawed at home before consumption. Dosage: At least 3 slices of bread 6 days per week for 16 weeks

SUMMARY:
This is a multicenter study testing the effect of bread containing beta-glucan on glycemic control in participants with intermediate hyperglycemia. The main hypothesis of the study is that bread enriched with beta-glucan will have a positive effect on blood glucose control (HbA1c) in persons with intermediate hyperglycemia.

Bread (intervention and control) will be produced by Nofima (Ås, Norway) using food-grade beta-glucan from oat and barley and shipped to the study centers (Bergen (N), Gothenburg (S), Paderborn, and Leipzig (D)) and there distributed for free to the participants of the study. The study will last for 16 weeks with measurements at baseline, after 8 weeks and after 16 weeks. Blood and urine samples will be taken, anthropometry and body composition measured, and questionnaires on health status and socio-economic status, physical activity, nicotine use, alcohol habits, chronotype, quality of life, and consumer acceptance of the study bread will be filled in.

DETAILED DESCRIPTION:
Carbohydrates are the main source of energy in most European countries with intakes ranging from 40-60% of total energy. Consequently, the role of its quality and quantity for the development of metabolic diseases is the focus of substantial debate. Notwithstanding, replacing processed carbohydrates with unprocessed carbohydrates is regarded as a major strategy to improve public health. This is to a substantial degree based on strong observational evidence that higher intakes of dietary fiber (cereal grains containing the same relative proportions of bran, germ, and endosperm as the intact caryopsis) are associated with lower risks of total mortality, cardiovascular morbidity, and mortality, type 2 diabetes mellitus (T2DM) incidence and cancer mortality. Nonetheless, data from medium- to long-term intervention studies among adults are less conclusive regarding the benefits of whole-grain consumption on glycemic control, bodyweight and serum lipids. In fact, benefits may be largely confined to whole grains stemming from oats or barley, calling for explicit consideration of these whole grains and/or its mechanistically relevant component.

Adding complexity, many commonly consumed whole grains or products rich in dietary fiber are characterized by a high glycemic index (GI>70), in fact, a high dietary fiber content will not predict a low glycemic response. The GI describes the glycemic potency of the available carbohydrates in a food, is measured under defined conditions and is used to calculate the glycemic load (GL: GI x amount of available carbohydrates). Preferred consumption of high GI grain products is of concern since a higher dietary GI and GL may be causally linked to a substantial increase in T2DM risk and may translate into a considerable health burden.

In European societies, T2DM prevalence is increasing as a result of higher overweight and obesity rates and increases in longevity. Efforts are hence needed to develop carbohydrate-based food items that are both rich in fiber and whole grain and have a low GI and tailored to the dietary habits of middle-aged adults with insulin resistance (also called 'pre-diabetes' or intermediate hyperglycemia defined by intermediately increased HbA1c levels). This stage precedes clinical T2DM and affects up to 30% of adults in Western societies.

Enrichment with selected fibers, e.g. beta-glucan from oat and barley, may offer an alternative to whole grain kernel breads, which may not meet consumer preferences and is also endorsed by EFSA health claims. Preliminary small-scale studies indicate acute, short- and longer-term benefits of such bread for glycemic and/or insulinemic responses among persons with T2DM or at risk of T2DM. However, these studies suffer, besides the small sample sizes, from high amounts of test food (8 servings per day = 320 g bread) and use of white bread as a comparator. The present study will test whether habitual consumption of a bread containing oat bran concentrate and meeting the high beta-glucan content of the EFSA claim (4.3 g beta-glucan per 30 g available carbohydrate) compared to normal wheat bread high in whole grain but without kernels will affect glycemic control over a period of 16 weeks.

Main hypothesis The main hypothesis of the study is that bread enriched with beta-glucan will have a positive effect on blood glucose control (HbA1c) in persons with intermediate hyperglycemia.

Objectives Main objective: Establish whether replacement of habitual bread intake with a low GI bread containing beta-glucan improves glycemic control among persons at risk for T2DM.

Secondary objectives: Examine the effects of the intervention on capillary blood glucose, body composition and serum lipid levels, and address consumer acceptance of the intervention bread.

Study procedures This is a multicenter study testing the effect of bread containing beta-glucan on glycemic control in participants with intermediate hyperglycemia.

Breads (intervention and control) will be produced by Nofima (Ås) using food-grade beta-glucan from oat and barley and shipped to the study centers (Bergen (N), Gothenburg (S), Paderborn and Leipzig (D)) and there distributed for free to the participants of the study. The study will last for 16 weeks with measurements at baseline, after 8 weeks and after 16 weeks. Blood and urine samples will be taken, anthropometry and body composition measured, and questionnaires on health status, chronotype, lifestyle, and acceptance of the breads will be filled in.

Recruitment of participants Each study site is responsible for the recruitment of the planned numbers of participants. Potential participants will be recruited through flyers and information to local General Practitioners, advertising in local newspapers, central and local social media announcements (websites of universities, Facebook). Potentially eligible participants will be invited to a screening visit and checked for eligibility and exclusion of undiagnosed 2TDM.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c 35-50 mmol/mol
* BMI ≥ 27 m2/kg
* regular bread eaters
* freezing capacity of at least 2 bread

Exclusion Criteria:

* chronic diseases like T2DM, CVD, cancer (within the last three years)
* unknown or untreated hypertension >160/100 mmHg
* celiac diseases, intolerance, or allergies for nuts, milk, eggs, wheat, mustard, seeds
* use of anti-diabetic drugs
* pregnancy and breastfeeding
* patients planned to have or had a bariatric surgery
* alcohol abuse

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 16 weeks
  Measurement of HbA1c

SECONDARY OUTCOMES:
fasting capillary blood glucose | 16 weeks
  Measurement of fasting capillary glucose
Body weight | 16 weeks
  Measurement of body weight
Lipids | 16 weeks
  Measurement of total cholesterol, LDL-C, HDL-C, triglycerides
Consumer acceptance | 8 weeks
  Questionnaire on consumer acceptance (scale 1-9, 9 indicates "tastes really good" or "very hungry")
Liver enzymes | 16 weeks
  Measurement of serum concentrations of ALAT (U/L) and ASAT (U/L)
Fecal Microbiota | 16 weeks
  Analyse the change in the composition of the fecal microbiota using 16S sequencing
Continuous blood glucose measurements | 1 week at baseline and after 16 weeks
  Measurement of Continuous blood glucose in a sub-population
Compliance | 16 weeks
  Compliance of the intervention/control will be evaluated using compliance journals and 24-hour recalls as the basis for sensitivity analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jutta Dierkes, PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hjorth T, Schadow A, Revheim I, Spielau U, Meyer K, Rieder A, Varela P, Ballance S, Koerner A, Landberg R, Buyken AE, Dierkes J, Rosendahl-Riise H. Effectiveness of regular oat beta-glucan-enriched bread compared with whole-grain wheat bread on long-term glycemic control in adults at risk of type 2 diabetes: a randomized controlled trial. Am J Clin Nutr. 2025 Sep;122(3):724-732. doi: 10.1016/j.ajcnut.2025.06.018. Epub 2025 Jun 24. PMID 40571100
- [Derived] Hjorth T, Schadow A, Revheim I, Spielau U, Thomassen LM, Meyer K, Piotrowski K, Rosendahl-Riise H, Rieder A, Varela P, Lysne V, Ballance S, Koerner A, Landberg R, Buyken A, Dierkes J. Sixteen-week multicentre randomised controlled trial to study the effect of the consumption of an oat beta-glucan-enriched bread versus a whole-grain wheat bread on glycaemic control among persons with pre-diabetes: a study protocol of the CarbHealth study. BMJ Open. 2022 Aug 23;12(8):e062066. doi: 10.1136/bmjopen-2022-062066. PMID 35998955